CLINICAL TRIAL: NCT06481501
Title: Mindfulness Intervention for Individuals With HIV and Chronic Pain
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources diverted to another project
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Adam Hanley, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00005157
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain; HIV Infections
MeSH Terms: conditions — Chronic Pain; HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ONE Mindfulness-Oriented Recovery Enhancement (Experimental): One MORE is a 2-hour adaptation of the manualized MORE program and will be divided into four, 30-minute segments. In the first segment, participants will be introduced to mindfulness and guided though a body scan practice, which directs participants to systematically shift attention from one part of the body to the next. Mindful pain management will be the focus of the second segment and participants will be guided through a mindfulness of pain practice in which they will learn to deconstruct pain into sensory, emotional, cognitive, and behavioral components. The third segment will focus on managing the negative thoughts and emotion that can amplify pain with mindful reappraisal, and the fourth segment will focus on increasing the positive emotions that can attenuate pain with mindful savoring.
  Interventions: Behavioral: ONE Mindfulness-Oriented Recovery Enhancement
- Treatment As Usual (No Intervention): In the Treatment as Usual (TAU) condition, participants will complete all study assessments (pre-treatment, post-treatment, 2-week, 4-week) without receiving any ONE MORE training. During their study involvement, TAU participants will be encouraged to continue any previously initiated treatment but discouraged from beginning any new form of treatment. Those in the TAU condition will not be sent any training materials.

INTERVENTIONS:
Behavioral: ONE Mindfulness-Oriented Recovery Enhancement — One MORE is a 2-hour adaptation of the manualized MORE program and will be divided into four, 30-minute segments. In the first segment, participants will be introduced to mindfulness and guided though a body scan practice, which directs participants to systematically shift attention from one part of the body to the next. Mindful pain management will be the focus of the second segment and participants will be guided through a mindfulness of pain practice in which they will learn to deconstruct pain into sensory, emotional, cognitive, and behavioral components. The third segment will focus on managing the negative thoughts and emotion that can amplify pain with mindful reappraisal, and the fourth segment will focus on increasing the positive emotions that can attenuate pain with mindful savoring.
  Arms: ONE Mindfulness-Oriented Recovery Enhancement

SUMMARY:
This project is a single-site, two-arm, randomized controlled pilot study examining the impact of a 2-hour version of Mindfulness-Oriented Recovery Enhancement (ONE MORE) training for individuals with HIV and chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic pain
* Be HIV+
* 18 years of age or older
* Fluent English speaker
* Will commit to try no other new treatments during study duration

Exclusion Criteria:

* Not having HIV
* Being unable to follow tasks due to pain level
* Prior mindfulness training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2026-07-25 (Estimated)

PRIMARY OUTCOMES:
Recruitment Feasibility | 4 months
  Examine recruitment rates during the 4 months of recruitment.
Intervention Adherence | 2 Hours
  Examine the percentage of participants completing their 2-hour intervention session.
Treatment Acceptability | Completed immediately after the 2-hour ONE MORE training
  Treatment acceptability will be assessed with a 12-item adaptation of the Treatment Framework of Acceptability questionnaire. Higher scores reflect greater acceptability.

SECONDARY OUTCOMES:
Global Impression of Change | Completed at 2- and 4-week follow-ups
  Treatment related improvement will be assessed with the Patient Global Impression of Change scale. Scores range from 0 to 7, with higher scores reflecting greater treatment related improvement.

OTHER OUTCOMES:
Acute Pain Unpleasantness | Will be completed immediately before and after the 2-hour intervention session
  Change in acute pain unpleasantness will be measured with an individual item ("How unpleasant is your pain, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain unpleasantness.
Acute Pain Intensity | Will be completed immediately before and after the 2-hour intervention session
  Change in acute pain intensity will be measured with an individual item ("How much pain do you have, right now?") rated on a numeric rating scale. Scores range from 0 to 10, with higher scores reflecting greater acute pain intensity.
Daily Pain Intensity | Daily for 4 weeks
  Change in daily pain intensity from from the first post-intervention day through the 4-week follow-up will be assessed with the pain intensity item from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain intensity.
Daily Pain Interference | Daily for 4 weeks
  Change in daily pain interference from from the first post-intervention day through the 4-week follow-up will be assessed with the two pain interference items from the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater pain interference.
Chronic Pain | Baseline, 2 weeks post-treatment, 4 week post-treatment]
  Change in chronic pain from baseline through 4-week follow-up will be assessed with the Pain, Enjoyment, and General Activity scale. Scores range from 0 to 10, with higher scores reflecting greater chronic pain.
Sleep | Baseline, 2 weeks post-treatment, 4 week post-treatment]
  Change in sleep from baseline through 4-week follow-up will be assessed with the PROMIS Sleep Disturbance Short Form. Scores range from 6 to 30, with higher scores reflecting worse sleep.
Pain Catastrophizing | Baseline, 2 weeks post-treatment, 4 week post-treatment
  Change in pain catastrophizing from baseline through 4-week follow-up will be assessed with the Pain Catastrophizing Scale. Scores range from 0 to 52, with higher scores reflecting greater pain catastrophizing.
Depression | Baseline, 2 weeks post-treatment, 4 week post-treatment]
  Change in depression from baseline through 6-week follow-up will be assessed with the Patient Health Questionnaire-2. Scores range from 0 to 6, with higher scores reflecting greater depression.
Anxiety | Baseline, 2 weeks post-treatment, 4 week post-treatment
  Change in anxiety from baseline through 4-week follow-up will be assessed with the Generalized Anxiety Disorder 2-item. Scores range from 0 to 6, with higher scores reflecting greater anxiety.
Prescription Pain Medication Use | Baseline, 2-weeks post-treatment, 4 weeks post-treatment
  Change in prescription pain medication misuse from baseline through 4-week follow-up will be assessed with the PROMIS Prescription Pain Medication Misuse Short Form. Scores range from 7 to 35, with higher scores reflecting greater medication misuse.
Substance Use | Baseline, 2-weeks post-treatment, 4 weeks post-treatment
  Change in substance misuse from baseline through 4-week follow-up will be assessed with the Severity of Substance Use Short Form 7a. Scores range from 7 to 35, with higher scores reflecting greater substance use
Alcohol Use | Baseline, 2-weeks post-treatment, 4 weeks post-treatment
  Change in alcohol use from baseline through 4-week follow-up will be assessed with the PROMIS v1.0 Alcohol Use - Short Form 7a. Scores range from 7 to 35, with higher scores reflecting greater alcohol use
Nicotine Use | Baseline, 2-weeks post-treatment, 4 weeks post-treatment
  Change in nicotine use from baseline through 4-week follow-up will be assessed with the Smoking: Nicotine Dependence for All Smokers - Short Form 4a. Scores range from 4 to 20, with higher scores reflecting greater nicotine use
Mindful Pain Management Mindful Pain Management | Baseline, 2 weeks post-treatment, 4 week post-treatment
  Change in the use of mindfulness for pain management from baseline through 4-week follow-up will be assessed with the Mindful Reappraisal of Pain Scale. Scores range from 0 to 54, with higher scores reflecting greater mindful pain management.
Self-Transcendent Experiences Self-Transcendent Experiences | Baseline, 2 weeks post-treatment, 4 week post-treatment
  Change in the the frequency of self-transcendent experiences from baseline through 4-week follow-up will be assessed with the Nondual Awareness Dimensional Assessment. Scores range from 0 to 5, with higher scores reflecting more frequent self-transcendent experiences.
Self Transcendent State | Will be completed immediately before and after the 2-hour intervention session
  Change in self-transcendent state from immediately before treatment to immediately after treatment will be assessed with the Nondual Awareness Dimensional Assessment- State Version. Scores range from 0 to 10, with higher scores reflecting deeper states of self-transcendence.
Trait-Like Decentering | Baseline, 2-weeks post-treatment, 4 weeks post-treatment
  Change in meta-awareness, non-reactivity, and acceptance from baseline through 4-week follow-up will be assessed with the Metacognitive Processes of Decentering Scale. Scores range from 15 to 75, with higher scores reflecting greater emotional balance
State-Like Decentering | Will be completed immediately before and after the 2-hour intervention session
  Change in decentering from immediately before treatment to immediately after treatment (i.e., 2 hours later) will be assessed with the Metacognitive Processes of Decentering Scale. Scores range from 0 to 10, with higher scores reflecting greater de-centering
Savoring Beliefs | Baseline, 2 weeks post-treatment, 4 week post-treatment
  Change in individuals' perceptions of their ability to derive pleasure through anticipating upcoming positive events, savoring positive moments, and reminiscing about past positive experiences were measured from baseline through 4-week follow-up will be assessed with the Savoring Beliefs Inventory. Scores range from 0 to 4, with higher scores reflecting stronger enjoyment of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Brain Science and Symptom Management Center, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No